CLINICAL TRIAL: NCT06782113
Title: Prospective Study on the Safety and Efficacy of the UNILEXA Exoskeleton for Regular Verticalization and Assisted Walking
Brief Title: Safety and Efficacy of the UNILEXA Exoskeleton for Regular Verticalization and Assisted Walking
Status: Active, not recruiting | Type: Observational
Sponsor: MEBSTER (Industry)
Responsible Party: Sponsor
Other Study IDs: 202411 J01
Record Dates: First submitted 2024-12-12; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injury; Exoskeleton Device
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The primary objective of this clinical follow-up is to analyze data regarding the safety of the UNILEXA passive exoskeleton post-market. The secondary objective is to assess the effectiveness of the device in improving activities of daily living (ADL) through improved mobility, endurance and health-related quality of life (QoL). The aim of this study is to provide real-world evidence to support wider clinical and home use of the exoskeleton. This observational study is designed for 6 participants from a population of individuals with lower limb paralysis. The study will have a duration of 14 weeks. During this period, participants will visit Janske Lazne three times for routine measurements in a biomechanical laboratory, which will be integrated into their usual physiotherapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with lower limb paralysis due to spinal cord injury (T5-T12 lesion) in chronic phase (> 6 months)
* Age 18 years and older.
* ASIA score: AIS A or AIS B.
* Ability to provide informed consent and follow study procedures.
* Weight below 100 kg.
* Height between 165 - 195 cm. (PI can decide to include participants outside of this range. The IFU specifies an EXTENDED range of 160 - 200 cm with certain conditions.)

Exclusion Criteria:

* Severe contractures in the lower limbs.
* Spasticity greater than 2 according to the Modified Ashworth Scale (MAS).
* Autonomic dysreflexia.
* Spinal instability.
* Untreated deep vein thrombosis.
* Untreated fractures of the pelvis or limbs.
* Advanced osteoporosis.
* Complete tetraplegia.
* Lack of upper limb control grade 3 or less, according to the ASIA test.
* History of fracture due to osteoporosis.
* Medication that increases the chance of fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with lower limb paralysis who have purchased and are actively using the UNILEXA exoskeleton.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events and Adverse Device Effects [Safety Assessment] | From enrollment to the end of observation at 14 weeks
  Analyze data regarding the safety of the UNILEXA exoskeleton by determining the incidence of adverse events (AEs) and adverse device effects (ADEs), such as falls, skin injuries, and other injuries, over the study period.

SECONDARY OUTCOMES:
Health-Related Quality of Life (QoL) | From enrollment to the end of observation at 14 weeks
  To assess improvements in health-related quality of life (QoL) using the WHOQOL-BREF questionnaire, a standardized questionnaire measuring QoL across four domains: physical, psychological, social relationships, and environment.
  Scale range: 0-100. Interpretation: Higher scores indicate better quality of life.
User Satisfaction Measured by QUEST 2.0 | From enrollment to the end of observation at 14 weeks
  To assess user satisfaction with the UNILEXA exoskeleton using the QUEST 2.0 questionnaire. This evaluates satisfaction with the device and associated services.
  QUEST 2.0: A validated user satisfaction questionnaire consisting of 12 items across two subscales: device satisfaction and service satisfaction. Each item is rated on a 5-point Likert scale (1 = not satisfied at all, 5 = very satisfied).
Time to Complete the 10-Meter Walk Test (10MWT) | From enrollment to the end of observation at 14 weeks
  To evaluate the time required to walk 10 meters at a comfortable speed.
  Unit of Measure: Seconds. Interpretation: Lower times indicate better functional mobility.
Time to Complete the Timed Up and Go (TUG) Test | From enrollment to the end of observation at 14 weeks
  To assess mobility performance by measuring the time required to stand up from a chair, walk 3 meters, turn, and return to sit in the chair.
  Unit of Measure: Seconds. Interpretation: Lower times indicate better functional mobility.
Level of Assistance Required for Mobility | From enrollment to the end of observation at 14 weeks
  To evaluate the level of physical assistance required during mobility tasks using a 6-point ordinal scale.
  Scale range: 0-5, where 0 = no assistance and 5 = full physical assistance required.
  Interpretation: Lower scores indicate better functional independence.
Rating of Perceived Exertion Measured by Borg RPE | From enrollment to the end of observation at 14 weeks
  To evaluate the perceived exertion of participants during mobility tasks using the Borg RPE scale.
  Borg RPE Scale: Measures exertion on a scale from 0-10, where 0 = no exertion and 10 = maximal exertion.
Pain Intensity Measured by Visual Analog Scale (VAS) | From enrollment to the end of observation at 14 weeks
  To assess the pain intensity experienced by participants during mobility tasks using the Visual Analog Scale (VAS).
  VAS Scale: Measures pain on a scale from 0-10, where 0 = no pain and 10 = the worst imaginable pain.
Cognitive and Physical Workload Measured by NASA-TLX | From enrollment to the end of observation at 14 weeks
  To evaluate the cognitive and physical workload experienced by participants during mobility tasks using the NASA Task Load Index (NASA-TLX) questionnaire.
  NASA-TLX: A multidimensional workload assessment tool with six subscales: mental demand, physical demand, temporal demand, performance, effort, and frustration.
  Scale range: 0-20 for each subscale. Interpretation: Higher scores indicate greater workload in each category.

OTHER OUTCOMES:
Amplitude of Vertical and Lateral Acromion Marker Movement | From enrollment to the end of observation at 14 weeks
  To assess compensatory movements by analyzing the amplitude of reflective markers placed on the acromion.
  Parameters measured: Amplitude of vertical and lateral movements. Units of Measure: Millimeters (mm). Data summarization: Mean and standard deviation of marker amplitude across all trials.
Amplitude of Pelvic Angular Movements (Rotation, Hiking, Tilting) | From enrollment to the end of observation at 14 weeks
  To evaluate biomechanical adaptations by measuring the amplitude of pelvic angular movements in three major planes:
  Pelvic Rotation: Angular displacement in the transverse plane. Pelvic Hiking: Angular displacement in the coronal plane. Pelvic Tilting: Angular displacement in the sagittal plane. Units of Measure: Degrees (°). Data summarization: Mean and standard deviation of angular displacement for each type of movement (rotation, hiking, tilting) across all trials.
Number of Steps Taken Per Training Session | From enrollment to the end of observation at 14 weeks
  To evaluate participant progress during the training phase by recording the number of steps taken in each training session.
  Unit of Measure: Number of steps. Data summarization: Total number of steps per session and average across all sessions.
Total Distance Walked Per Training Session | From enrollment to the end of observation at 14 weeks
  To assess participant mobility during the training phase by measuring the total distance walked in each training session.
  Unit of Measure: Meters (m). Data summarization: Total distance walked per session and average across all sessions.
Duration of Use Per Training Session | From enrollment to the end of observation at 14 weeks
  To assess participant endurance during the training phase by recording the duration of each training session.
  Unit of Measure: Minutes. Data summarization: Total duration per session and average across all sessions.
Heart Rate During Laboratory Tests | From enrollment to the end of observation at 14 weeks
  To assess physiological responses during training sessions by measuring participants' heart rates.
  Unit of Measure: Beats per minute (BPM). Data summarization: Average heart rate during each session and across all sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Státní léčebné lázně Janské Lázně, státní podnik, Janske Lazne, Czechia